CLINICAL TRIAL: NCT06874959
Title: A Randomized Control Trail: Evaluation of the Pain Relief Effect of Battlefield Acupuncture on Patients With Chronic Low Back Pain Due to Lumbar Spine Degeneration.
Brief Title: Evaluation of the Pain Relief Effect of Battlefield Acupuncture on Patients With Chronic Low Back Pain Due to Lumbar Spine Degeneration.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Medicine and Pharmacy at Ho Chi Minh City (Other)
Responsible Party: Principal Investigator, Bui Pham Minh Man, Doctor of Philosophy, University of Medicine and Pharmacy at Ho Chi Minh City
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2469/DHYD-HDDD
Record Dates: First submitted 2025-02-26; First posted 2025-03-13 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Spondylosis Lumbar
Keywords: Lumbarsacral Spondylosis; Battlefield acupuncture; Ear acupuncture; Low back pain
MeSH Terms: conditions — Spondylosis; Low Back Pain | interventions — Acupuncture, Ear; Acetaminophen

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experiment (Experimental): Auricular acupuncture + Electro acupuncture + Pain medication
  Interventions: Device: Ear acupuncture; Device: Electro-acupuncture; Drug: Paracetamol 500 mg
- Sham Comparator (Sham Comparator): Sham ear acupuncture + Electro acupuncture + Pain medication
  Interventions: Device: Electro-acupuncture; Drug: Paracetamol 500 mg; Device: Sham ear acupuncture

INTERVENTIONS:
Device: Ear acupuncture — (According to the guidelines provided in the "BFA - Acupuncture Manual" of the USAF Center for Integrative and Complementary Medicine.)
  Procedure:
  * Practitioner: Traditional medicine doctor with a practicing certificate.
  * Tools: Khanh Phong auricular acupuncture needles (license: 287/BYTYDCT)
  * Before needling: Disinfect the skin on both outer ears.
  * Insertion depth: Auricular needles penetrate the skin to a depth of 1.3 mm. Insert the auricular needles alternately on the right and left sides at the following acupoints: Cingulate gyrus, Subcortex, Omega 2, Shen Men, and Zero point. The insertion process stops when one of the following three criteria is met: (1) The patient experiences a 40% reduction in pain on the Visual Analog Scale (VAS), (2) The patient refuses to continue the insertion, or (3) A total of 10 needles have been inserted.
  * After needling: Patient may feel slight pain in the ear area or de qi (a sensation of aching, warmth, and redness at the needling site).
  Arms: Experiment
Device: Electro-acupuncture — According to the "Guidelines for the Diagnosis and Treatment of Diseases by Traditional Medicine, combining Traditional Medicine with Modern Medicine" - 2020 - Ministry of Health of Viet Nam.
  Procedure:
  * Practitioner: Traditional medicine doctor with a practicing certificate.
  * Tools: Khánh Phong ARLO acupuncture needles, size 0.3 x 25 mm (lincense: TKHQ:102664344900)
  * Disinfect the lumbar region skin.
  * Needle insertion: Insert needles perpendicular to the patient's skin, to a depth of 20 mm. Location: Dai truong du (BL25), Than du (BL23), Jiaji at L4-L5, L5-S1 (Ex-B2), Uy trung (BL40), Yeu duong quan (GV3). After insertion, attach the electrode clips to the needle ends.
  * Electric stimulation: Use a current of 100Hz for 20 minutes - mixed wave.
  * Post-needling: Patient may feel a sensation of de qi (aching, warmth, and redness at the needling site).
Drug: Paracetamol 500 mg — According to the "Guidelines for the Diagnosis and Treatment of Diseases by Traditional Medicine, combining Traditional Medicine with Modern Medicine" - 2020 - Ministry of Health of Viet Nam.
  * Prescriber: Traditional medicine doctor with a practicing certificate.
  * Paracetamol 500mg x 9 tablets: Take 1 tablet per dose, to be used when the pain score on the Visual Analog Scale (VAS) is ≥ 30mm, not exceeding 6 tablets/day. (If the patient still has medication from the previous visit, only prescribe the total amount needed to make up 9 tablets).
Device: Sham ear acupuncture — Study uses patches with non-skin-penetrating cotton, at the intervention acupoint areas. Using acupoints matching with the intervention group helps reduce the patients' ability to predict their study group, and the non-penetrating and non-rotating cotton ensure that there is no analgesic effect on the lumbar area caused by auriculotherapy.
  Acupoint location: Cingulate gyrus, Subcortex, Omega 2, Shen Men, and Zero points
  Arms: Sham Comparator

SUMMARY:
The Global Burden of Disease's 2023 study shows that lower back pain affects over 619 million people worldwide, with projections reaching 843 million by 2050. It is a common symptom of lumbar spine degeneration, with 84.2% of patients experiencing it. To address this issue, Vietnam's Ministry of Health has released guidelines on "Lumbar Spine Pain" (Yêu thống), combining traditional and modern medicine, including acupuncture, to alleviate pain. However, to achieve better treatment outcomes, the combination of multiple interventions, such as different types of acupuncture, is required. Additionally, the USAF's Integrative Medicine and Acupuncture Center released guidelines in 2021 for Battlefield Acupuncture (BFA), a rapid, safe, and effective pain relief method. Internationally, there are studies on BFA for various types of pain, including lower back pain, but none in Vietnam. Therefore, the investigators conducted this study to evaluate the effects of BFA combined with electroacupuncture and pain medication on chronic lower back pain patients with lumbar spine degeneration in Vietnam.

DETAILED DESCRIPTION:
The Global Burden of Disease's 2023 study shows that lower back pain affects over 619 million people worldwide, with projections reaching 843 million by 2050. It is a common symptom of lumbar spine degeneration, with 84.2% of patients experiencing it. To address this issue, Vietnam's Ministry of Health has released guidelines on "Lumbar Spine Pain" (Yêu thống), combining traditional and modern medicine, including acupuncture, to alleviate pain. However, to achieve better treatment outcomes, the combination of multiple interventions, such as different types of acupuncture, is required. Additionally, the USAF Integrative Medicine and Acupuncture Center published a guideline in 2021 for BFA ear acupuncture, specifying points to be acupunctured in the following order: Cingulate gyrus, Subcortex, Omega 2, Shen Men, and Zero. Currently, this method has been extensively researched and has shown its potential in both acute and chronic pain, such as chronic musculoskeletal pain in cancer patients, acute back pain in intensive care units, and non-specific chronic back pain. Despite the proven effectiveness in many studies and the publication of detailed guidelines for BFA in the USA, this potential pain relief method has not been evaluated for effectiveness in Vietnam. Therefore, the investigators conducted this study to evaluate the effects of BFA combined with electroacupuncture and pain medication on chronic lower back pain patients with lumbar spine degeneration in Vietnam.

The investigators conduct a single blind randomized control trail, from March 2025 to October 2025, on 60 low-back-pain patients diagnosed with lumbar spine degeneration (or lumbosacral spondylosis). These patients will be randomly divided into two groups: A (intervention group - 30 patients) and B (sham group - 30 patients). The patients in group A will receive ear acupuncture, while the patients in group B will receive sham ear acupuncture. All patients will be treated with electroacupuncture and prescribed pain medication. Each patient will undergo a 10-day course of treatment (3 sessions per week, each session 1 day apart from the previous one). The details of the intervention will be discussed further below. At the end of each session, the investigators will collect Visual Analog Scale (VAS) scores, and the number of pain medications used. At the end of the 5th and the 10th session, the investigators will collect Brief Pain Inventory (BPI) scores.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 20 years and older.
* Patients diagnosed with lumbar spine degeneration (Imaging and clinical criteria according to the "Guidelines for Diagnosis and Treatment of Musculoskeletal Diseases" - Ministry of Health of Viet Nam 2014; AAFP-2024).
* Patients with back pain with a VAS score of ≥ 50mm, continuous or recurrent with the same initial diagnosed cause, lasting from the time of initial diagnosis to the time of study participation for ≥ 3 months.
* Individuals who have never used auricular acupuncture.
* Voluntarily agree to participate in the study.

Exclusion Criteria:

* Individuals with cognitive disorders (Glasgow < 13 points).
* Individuals are allergic to any component of the ear acupressure seeds, or experiencing anxiety, fear of needles, or with a history of acupuncture syncope.
* Patients with symptoms of saddle anesthesia, urinary or fecal incontinence, paresthesia or muscle atrophy, progressive muscle weakness.
* History of cancer or currently undergoing cancer treatment, or unexplained weight loss.
* Patients who are awakened at night due to back pain.
* Patients contraindicated the medication used in the study: paracetamol.
* Pregnant or breastfeeding women.
* Patients are currently experiencing systemic infection.
* Individuals with unhealed wounds, ear or lumbar region infections.
* Currently participating in an intervention study with another drug or device.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2025-03-15 (Actual); Primary Completion 2025-07-31 (Actual); Study Completion 2025-08-31 (Actual)

PRIMARY OUTCOMES:
Visual Analog Scale | Baseline, during procedure
  The Visual analog scale is a continuous scale consisting of a horizontal line (HVAS) or a vertical line (VVAS), typically 10 cm (100 mm) in length. The scale is usually anchored at both ends with the descriptors "no pain" (score 0) and "worst imaginable pain" (score 100 [100 mm scale]). To avoid clustering scores around a preferred number, intermediate points should not be numbered or verbally described. The timing of data collection varies between different studies or examinations, but most respondents are asked to report pain intensity "currently" or pain intensity "in the past 24 hours."
Brief Pain inventory | Baseline, session 1st, session 5th, session 10th
  The BPI is a self-assessment scale for sensory aspects and responses to pain. The scale includes two parts: pain intensity and the degree of impact on various aspects of life. The impact is assessed in different areas of daily living such as sleep, mobility, and emotional well-being. The survey period can be either 7 days or 24 hours. IMMPACT (Initiative on Methods, Measurement, and Pain Assessment in Clinical Trials) recommends that BPI be used for clinical trials with patients suffering from chronic pain.
  BPI begins with a screening question about the location of the pain that the patient feels needs attention. The main sections include pain intensity scale and the impact of pain. A numerical rating scale from 0 to 10 is used for all items. The endpoints for the pain intensity scale are 0 = 'no pain' and 10 = 'pain as bad as you can imagine', while the endpoints for the quality-of-life scale are 0 = 'no impact' and 10 = 'total impact'.
Pain medication used | During procedure
  The use of pain medications serves as an indicator of the efficacy of acupuncture as a pain-relief intervention. An increased dependence on analgesic medications among patients signifies a diminished therapeutic effect of acupuncture in alleviating pain symptoms.

CONTACTS AND LOCATIONS:
Locations (2):
- Vietnam (2):
  - Traditional Chinese Medicine faculty - Thống Nhất Hospital, Ho Chi Minh City
  - University medical center HCMC branch 3, Ho Chi Minh City

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Song CY, Chen CH, Chen TW, Chiang HY, Hsieh CL. Assessment of Low Back Pain: Reliability and Minimal Detectable Change of the Brief Pain Inventory. Am J Occup Ther. 2022 May 1;76(3):7603205040. doi: 10.5014/ajot.2022.044420. PMID 35301518
- [Background] Hawker GA, Mian S, Kendzerska T, French M. Measures of adult pain: Visual Analog Scale for Pain (VAS Pain), Numeric Rating Scale for Pain (NRS Pain), McGill Pain Questionnaire (MPQ), Short-Form McGill Pain Questionnaire (SF-MPQ), Chronic Pain Grade Scale (CPGS), Short Form-36 Bodily Pain Scale (SF-36 BPS), and Measure of Intermittent and Constant Osteoarthritis Pain (ICOAP). Arthritis Care Res (Hoboken). 2011 Nov;63 Suppl 11:S240-52. doi: 10.1002/acr.20543. No abstract available. PMID 22588748
- [Background] Bielewicz J, Daniluk B, Kamieniak P. VAS and NRS, Same or Different? Are Visual Analog Scale Values and Numerical Rating Scale Equally Viable Tools for Assessing Patients after Microdiscectomy? Pain Res Manag. 2022 Mar 29;2022:5337483. doi: 10.1155/2022/5337483. eCollection 2022. PMID 35391853
- [Background] Murakami M, Fox L, Dijkers MP. Ear Acupuncture for Immediate Pain Relief-A Systematic Review and Meta-Analysis of Randomized Controlled Trials. Pain Med. 2017 Mar 1;18(3):551-564. doi: 10.1093/pm/pnw215. PMID 28395101
- [Background] Matz PG, Meagher RJ, Lamer T, Tontz WL Jr, Annaswamy TM, Cassidy RC, Cho CH, Dougherty P, Easa JE, Enix DE, Gunnoe BA, Jallo J, Julien TD, Maserati MB, Nucci RC, O'Toole JE, Rosolowski K, Sembrano JN, Villavicencio AT, Witt JP. Guideline summary review: An evidence-based clinical guideline for the diagnosis and treatment of degenerative lumbar spondylolisthesis. Spine J. 2016 Mar;16(3):439-48. doi: 10.1016/j.spinee.2015.11.055. Epub 2015 Dec 8. PMID 26681351
- [Background] Fox LM, Murakami M, Danesh H, Manini AF. Battlefield acupuncture to treat low back pain in the emergency department. Am J Emerg Med. 2018 Jun;36(6):1045-1048. doi: 10.1016/j.ajem.2018.02.038. Epub 2018 Feb 27. PMID 29550099
- [Background] Mao JJ, Liou KT, Baser RE, Bao T, Panageas KS, Romero SAD, Li QS, Gallagher RM, Kantoff PW. Effectiveness of Electroacupuncture or Auricular Acupuncture vs Usual Care for Chronic Musculoskeletal Pain Among Cancer Survivors: The PEACE Randomized Clinical Trial. JAMA Oncol. 2021 May 1;7(5):720-727. doi: 10.1001/jamaoncol.2021.0310. PMID 33734288
- [Background] Hướng dẫn Chẩn đoán và Điều trị bệnh theo Y học cổ truyền, kết hợp Y học cổ truyền với Y học hiện đại (2020).
- [Background] GBD 2021 Low Back Pain Collaborators. Global, regional, and national burden of low back pain, 1990-2020, its attributable risk factors, and projections to 2050: a systematic analysis of the Global Burden of Disease Study 2021. Lancet Rheumatol. 2023 May 22;5(6):e316-e329. doi: 10.1016/S2665-9913(23)00098-X. eCollection 2023 Jun. PMID 37273833